The Effect and Mechanism of Self-compassion on Reducing Materialism: A Randomized Controlled Trial of an Online Self-Compassion Intervention

ID (IRB Number): 202206260077

The Date of the Document: March 12, 2024

## The Effect and Mechanism of Self-compassion on Reducing Materialism: A Randomized Controlled Trial of an Online Self-Compassion Intervention Study protocol

The current study provided an initial investigation of the effect of self-compassion on reducing materialism and explored the basic psychological needs and self-esteem as potential mechanisms. Two studies would be conducted. Study 1 explored the relationships among variables with cross-sectional data, to explore the relationship between self-compassion and materialism, and test the mediating role of basic psychological needs and self-esteem. Study 2 developed a new online self-help self-compassion intervention and conducted a randomized control trial (i.e., intervention group and waitlist group) to further explore the casual effect of self-compassion on materialism, with the mediating effect of basic psychological needs and self-esteem.

## Study 1

Study 1 is a cross sectional study to explore the relationships between variables with natural daily data.

**Participants:** A total of 394 participants were recruited from websites. The inclusion criteria was having no current or previous mental disorder diagnosis. And only the participants who agree with the informed consent can continue to fill in the questionnaire.

*Measures:* The Chinese Version of Self-compassion Scale (SCS-C; Chen et al., 2011) was used to measure the self-compassion level of participants. The

Rosenberg Self-Esteem Scale (RSES; Rosenberg, 1965) was used to measure self-esteem using 10 items. The Balanced Measure of Psychological Needs Scale (BMPN; Sheldon & Hilpert, 2012) was used to measure basic psychological needs. The Material Tendencies Scale (MTS; Zhang & Xiao, 2019) was used to measure

**Data collection and analysis:** the data would be analysed by SPSS 26.0 and Mplus. In order to expore the relationship between variables, the correlation of variables would be conducted with SPSS 26.0. Additionly, mediation effect was analyzed by Mplus.

Expected results: (1) self-compassion was significantly correlated with materialism, and positively correlated with basic psychological needs, self-esteem; (2) the mediating effect of basic psychological needs and self-esteem would be supported, and the pathway from basic psychological needs to self-esteem would also be supported.

*Time plan:* Recruiting and filling out the questionnaires: November 1, 2020 to November 15, 2020

## Study 2

materialism.

Study 2 was an interventional study, and we conducted a randomized control trial (i.e., intervention group and waitlist group) to test the casual relationship between self-compassion and materialism, and the mediating role of basic psychological needs and self-esteem.

Participants: 381 participants registered for the study, and 309 met the

inclusion criteria, who filled the pretest. And participants would be randomly assigned

to intervention group (n = 154) or waitlist group (n = 155). The inclusion criteria were

as follows: (1) consented to accept randomization, finish the intervention and fill out

questionnaires and (2) had no current or previous mental disorder diagnosis.

*Measures:* the measurement used in study 2 were consistent with study 1.

Data collection and analysis: the data would be analysed with SPSS 26.0 and

Mplus. 2 (conditions) × 2 (times) ANOVAs were conducted to test the effect of the

intervention. The mediation effect was analyzed by Mplus to test the mediating role of

self-esteem, basic psychological needs and self-esteem.

Expected results: (1) compared with waitlist, the intervention could

significantly enhance self-compassion, self-esteem, basic psychological needs, and

decrease materialism; (2) the change of self-compassion mediates the group and all

other variables; (3) there would exist three mediating ways from self-compassion to

materialism: basic psychological needs, self-esteem, and the pathway from basic

psychological needs to self-esteem.

Time plan:

Recruiting: December 14, 2020 to December 20, 2020

Pretest: December 24, 2020 to December 29, 2020

Intervention conducted: January 4, 2021 to January 17, 2021

Posttest: January 25, 2021 to January 31, 2021

Follow up test: March 8, 2021 to March 14, 2021